CLINICAL TRIAL: NCT01733628
Title: Evaluation Study of Hypertension as a Predictor of Efficacy Bevacizumab (BV) in Combination With Chemotherapy (CT) in Metastatic Colorectal Cancer (MCC) and Metastatic Breast Cancer (MBC).
Brief Title: Evaluation of Hypertension as a Predictor of Efficacy Bevacizumab in Metastatic Breast Cancer and Colorectal Cancer
Acronym: BRECOL
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2011-04; GEI-BEV-2011-02 (Other: AEMPS)
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Breast Cancer
Keywords: Hypertension; Bevacizumab Response Predictors; Metastatic Breast Cancer; Metastatic Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Hypertension; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum or plasma) Tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bevacizumab + Chemotherapy: Patients who received the addition of Bevacizumab (BV) every 2-3 weeks to Chemotherapy (CT) with either oxaliplatin or irinotecan plus fluoropyrimidines in patients with Metastatic Colorectal Cancer (MCRC), either paclitaxel or capecitabine in patients with Metastatic Breast Cancer (MBC), as first-line therapy.

SUMMARY:
This is a multicenter, post-authorization observational with prospective follow-up (EPA-SP) study. Will be involved 137 metastatic breast cancer patients or metastatic colorectal cancer. The hypertension will be evaluated as a predictor of efficacy of bevacizumab associated with chemotherapy, in terms of progression-free survival (PFS) (Main endpoint).

The duration of the study will be approximately 42 months.

DETAILED DESCRIPTION:
Hypertension (HT) is the most common side effect seen in trials of bevacizumab in combination with chemotherapy. Based on the hypothesis that the development of hypertension during treatment would be an indicative of the successful blockade of the Vascular Endothelial Growth Factor (VEGF) pathway, different studies have explored retrospectively the relationship between hypertension and the results of treatment with bevacizumab.

This study aims to demonstrate the association between hypertension (diagnosed optimally) with efficacy to treatment with bevacizumab prospectively and secondly verify if blood pressure measures taken at home are a reflection of a diagnosis of hypertension.

Also have been explored different molecular markers involved in the pathway of VEGF which might be used as predictors of response. Therefore, this study includes the collection of blood samples (serum or plasma) and tumor tissue of patients included in this study, with the aim of exploring biomarkers that correlate with treatment efficacy and toxicity.

The diagnosis of hypertension (HT) will be performed using a Holter recording, and standard blood pressure footage will be collected during the first three cycles of treatment given the Common Toxicity Criteria of the National Cancer Institute-NCI CTCAE version 4.0 and the guidelines of the European Society of Cardiology and Hypertension, 2007.

Will be collected a sample of primary tumor and blood for patients who previously have consented it. Samples will be sent to a central laboratory for analysis of biomarkers.

An interim analysis will be conducted to assess the true incidence of hypertension. Based on this analysis, will be evaluated the need to recalculate the sample size.

At the end of the study, will be performed an analysis of correlation of data measured by standard BP (Blood Pressure) and Holter recording footage with the PFS. Moreover will be determined in serum, plasma and tumor tissue and certain biomarkers to correlate with efficacy to treatment with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

May only participate in the study patients (women and men) who meet all the following criteria:

1. MCC or MBC patients with chemotherapy and bevacizumab established indication. The first line systemic treatment planned for patients with MCC should be based in combination chemotherapy (oxaliplatin / irinotecan plus fluoropyrimidine) associated with bevacizumab. The first line systemic treatment planned for MBC patients should be based on a combination of paclitaxel or capecitabine plus bevacizumab.
2. Presence of measurable or evaluable disease according to RECIST 1.1, for the evaluation of the response to treatment.
3. Equal or more than 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Signed written informed consent.
6. Women of childbearing potential must have a negative pregnancy test in serum or urine conducted in the 7 days prior to the administration of chemotherapeutic treatment assigned by your doctor, and accept the use of double barrier contraception during the study (Note : Patients who are not of childbearing age may participate without using contraceptives. Women who are of childbearing age are those who: 1) have reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) within postmenopausal interval as determined by the laboratory, or 12 months of spontaneous amenorrhea), 2) have undergone bilateral oophorectomy with or without hysterectomy 6 weeks before, or 3) have undergone bilateral tubal ligation). Men also should use an adequate contraception method.

Exclusion Criteria:

Patients meeting any of the following circumstances will be excluded from the study:

1. Have received prior systemic anticancer therapy with chemotherapy for advanced disease or prior treatment with bevacizumab.
2. Treatment with an investigational agent or biological agent within 30 days prior to inclusion in the study.
3. Contraindications to treatment with chemotherapy and bevacizumab according to summary products characteristics.
4. Background or current history (within five years before the start of treatment) of other malignancies, except for colorectal carcinoma and breast cancer (patients with basal cell carcinoma or squamous cell skin or cervical carcinoma in situ treated curative may be included in the study).
5. Life expectancy less than 3 months.
6. Patients who are pregnant or breastfeeding.
7. Patients with an inadequate organ function (bone marrow, kidney and liver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic (disseminated at the time of diagnosis) breast cancer or colorectal cancer, treated with bevacizumab.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario de Elche
Locations (10):
- Spain (10):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Complejo Hospitalario Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - Centro Oncológico MD Anderson, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Rodriguez-Lescure A, Gallego J, Garcia-Alfonso P, Massuti B, Marquez R, Calvo L, Sanchez-Rovira P, Anton A, Chacon JI, Ciruelos E, Ponce JJ, Santaballa A, Valladares-Ayerbes M, Duenas MR, Alonso V, Aparicio J, Encinas S, Robles L, Escudero MJ, Caballero R, Bezares S, Garcia-Ortiz MV, Morales-Ruiz T, de la Haba-Rodriguez J. Hypertension as predictive factor for bevacizumab-containing first-line therapy in metastatic breast and colorectal cancer in BRECOL (GEICAM/2011-04) study. Clin Transl Oncol. 2024 Aug;26(8):1896-1907. doi: 10.1007/s12094-024-03411-w. Epub 2024 Apr 5. PMID 38578537
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2012 to July 2016, 143 patients were included.
Period: Overall Study
Arm/Group | Bevacizumab + Chemotherapy
Started | 143
Completed | 143
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 143
Age, Continuous [Median (Full Range); unit: years] | 61.18 [32.57 to 85.32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 143
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 67
    ECOG 1 | 72
    Unknown | 4
Blood Pressure Systolic [Mean (Full Range); unit: mmHg] | 129.4 [80 to 216]
Blood Pressure Diastolic [Mean (Full Range); unit: mmHg] | 74.73 [50 to 121]
Pulse [Mean (Full Range); unit: bpm] | 78.92 [52 to 128]
Women Menopausal Status [Count of Participants; unit: Participants] — Population: Only women were assessed for this measure
  Participants
    number analyzed (Participants) | 102
    Postmenopausal women | 75
    Premenopausal women | 27
Previous arterial hypertension [Count of Participants; unit: Participants]
  Previous arterial hypertension | 43
  No Previous arterial hypertension | 70
  Unknown | 30
Cancer type [Count of Participants; unit: Participants]
  Metastatic Colorectal Cancer (MCRC) | 65
  Metastatic Breast Cancer (MBC) | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With or Without Blood Pressure Increase as a Predictor of Progression Free Survival (PFS)
Description: The incidence of hypertension was studied during treatment with bevacizumab combined with chemotherapy. A Cox regression analysis was performed, entering as a dependent variable the PFS and as independent variable the Arterial Hypertension (AHT) (yes/no). AHT is introduced in the model of Cox as a time-dependent variable since its situation can change as length of the study. The date on which the AHT changes (passes from normotensive to hypertensive).
Time Frame: Up to 3 years
Population: There were 30 patients who were not included in Population per Protocol because of the following: 6 patients didn't fulfil inclusion and exclusion criteria, 8 patients didn't received Bevacizumab, 16 patients didn't have Holter assessment performed at baseline and/or at any other study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 113
Participants
  No AHT : 0 to 0.5 years | 19
  No AHT : 0.5 to 1 years | 11
  No AHT : 1 to 1.5 years | 6
  No AHT : 1.5 to 2 years | 4
  No AHT : 2 to 2.5 years | 1
  No AHT: 2.5 to 3 years | 1
  Yes AHT: 0 to 0.5 years | 94
  Yes AHT: 0.5 to 1 years | 58
  Yes AHT: 1 to 1.5 years | 25
  Yes AHT: 1.5 to 2 years | 13
  Yes AHT: 2 to 2.5 years | 7
  Yes AHT: 2.5 to 3 years | 5
Statistical Analysis 1: Comparison: Bevacizumab + Chemotherapy; Test type: Other — Type of statistical Test: Inequality; p = 0.8166, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.56 to 1.59]

2. Primary Outcome: Progression Free Survival (PFS)
Description: The PFS is the time from the patient receiving the first dose of chemotherapy for advanced disease to the date of progression, the administration of a new antineoplastic treatment that does not contain bevacizumab or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 113
Months | 10.19 (8.77)

3. Secondary Outcome: Number of Participants With "White Coat" AHT While at Home
Description: The incidence of "white coat" arterial hypertension (AHT) was evaluated comparing each of the measurements in medical attention (in a doctor office) with the measurement that was made at home (without a doctor).
  White Coat Hypertension is a phenomenon in which people exhibit a blood pressure level above the normal range, in a clinical setting, though they do not exhibit it in other settings.
Time Frame: Cycle 1, cycle 2, and cycle 3, up to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 113
Participants
  White coat AHT in cycle 1: No AHT | 60
  White coat AHT in cycle 1: Yes AHT | 6
  White coat AHT in cycle 1: Missing | 47
  White coat AHT in cycle 2: No AHT | 73
  White coat AHT in cycle 2: Yes AHT | 10
  White coat AHT in cycle 2: Missing | 30
  White coat AHT in cycle 3: No AHT | 65
  White coat AHT in cycle 3: Yes AHT | 6
  White coat AHT in cycle 3: Missing | 42

4. Secondary Outcome: Number of Participants With "White Coat" AHT With 24 Hours Ambulatory BP Measure
Description: The incidence of "white coat" arterial hypertension (AHT) was evaluated comparing each of the measurements with the measurement that was made in the hospital. Ambulatory Blood Pressure Monitoring (ABPM) is when the blood pressure is being measured as patient moves around, living her normal daily life.
  White Coat Hypertension is a phenomenon in which people exhibit a blood pressure level above the normal range, in a clinical setting, though they do not exhibit it in other settings.
Time Frame: Baseline, cycle 1, cycle 2, and cycle 3, up to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 113
Participants
  White coat AHT in baseline: No AHT | 94
  White coat AHT in baseline: Yes AHT | 14
  White coat AHT in baseline: Missing | 5
  White coat AHT in cycle 1: No AHT | 66
  White coat AHT in cycle 1: Yes AHT | 5
  White coat AHT in cycle 1: Missing | 42
  White coat AHT in cycle 2: No AHT | 83
  White coat AHT in cycle 2: Yes AHT | 9
  White coat AHT in cycle 2: Missing | 21
  White coat AHT in cycle 3: No AHT | 70
  White coat AHT in cycle 3: Yes AHT | 5
  White coat AHT in cycle 3: Missing | 38

ADVERSE EVENTS:
Time Frame: All adverse events occurred during the treatment and up to 30 days after the last dose were notified. All Serious Adverse Events (SAEs) that occurred within the first 3 cycles were recorded in the electronic Case Report Form (eCRF). Only those Grade 3-4 adverse events that were related to the treatment that occurred during the first 3 treatment cycles were recorded in the eCRF.
Description: The Safety Population (SP) included 135 patients who signed the Informed Consent and received at least 1 dose of Chemotherapy combined with Bevacizumab.
  The Intent to Treat (ITT) Population included 143 patients who signed the Informed Consent.
  Serious Adverse Events and/or Other (Not Including Serious) Adverse Events (AEs) have been calculated in the SP (n=135), and All-Cause Mortality have been calculated in the ITT population (n=143) as per protocol.
Groups:
- Bevacizumab + Chemotherapy: The Safety Population (SP) included 135 patients who signed the Informed Consent and received at least 1 dose of Chemotherapy combined with Bevacizumab.
  The Intent to Treat (ITT) Population included 143 patients who signed the Informed Consent.
  Serious Adverse Events and/or Other (Not Including Serious) Adverse Events (AEs) have been calculated in the SP (n=135), and All-Cause Mortality have been calculated in the ITT population (n=143).
Arm/Group | Bevacizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 9/143
Serious Adverse Events (participants affected / at risk) | 22/135
Other Adverse Events (participants affected / at risk) | 57/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=135)
Acute coronary syndrome (Cardiac disorders) | 1
Back pain (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
ICTUS (Cardiac disorders) | 1
Skin infection: Cellulitis (Infections and infestations) | 1
Lynph Gland Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Penile infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 2
Coronary Angiography (Surgical and medical procedures) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Neutrophil count decreased (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=135)
GGT increased (Investigations) | 8 — Grade 3
Hypertension (Cardiac disorders) | 11 — Grade 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 12 — Grade 3
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 3 — Grade 4
APTT increased (Investigations) | 3 — Grade 3
Abdominal pain (Gastrointestinal disorders) | 3 — Grade 3
Alanine aminotransferase increased (Investigations) | 1 — Grade 3
Anorexia (Nervous system disorders) | 1 — Grade 3
Aspartate aminotransferase increased (Investigations) | 1 — Grade 3
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 — Grade 3
Dehydration (General disorders) | 1 — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 — Grade 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 4
Fatigue (General disorders) | 3 — Grade 3
Diverticulitis (Gastrointestinal disorders) | 1 — Grade 3
Hyperkalemia (Investigations) | 1 — Grade 3
Hyponatremia (Investigations) | 1 — Grade 3
Fistulized perianal abscess (Gastrointestinal disorders) | 1 — Grade 3
LDL Cholesterol increased (Metabolism and nutrition disorders) | 3 — Grade 3
Lymphopenia (Blood and lymphatic system disorders) | 1 — Grade 3
Lymphopenia (Blood and lymphatic system disorders) | 2 — Grade 4
Mucositis oral (Gastrointestinal disorders) | 2 — Grade 3
Nausea (Gastrointestinal disorders) | 1 — Grade 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 — Grade 3
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2012-02-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT01733628/Prot_000.pdf